CLINICAL TRIAL: NCT05433818
Title: The Effect of Breastfeeding Education and Skin-to-Skin Contact on Breastfeeding Efficiency and Maternal Attachment: A Randomized Controlled Study
Brief Title: The Effect of Breastfeeding Education and Skin-to-Skin Contact on Breastfeeding Efficiency and Maternal Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-41997688-050.99-26938
Record Dates: First submitted 2022-06-13; First posted 2022-06-27 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-06

CONDITIONS: Breastfeeding; Postpartum; Infant Development
Keywords: Breastfeeding education; Breastfeeding efficiency; Infant; Maternal attachment; Skin-to-skin contact
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Skin-to-skin care (Experimental): Pregnant women will assigned to SSC were inform about SSC. SSC will ensured postpartum in a supported diagonal-flexion position continuously by the researchers for 45-120 minutes. Mothers in group A also benefit from the hospital's routine breastfeeding education service.
  As a result, after the SSC application, the mother will be evaluated with the breastfeeding efficiency scale and the maternal attachment scale.
  Interventions: Behavioral: Group A
- Breastfeeding Education (Active Comparator): Group B will received face-to-face breastfeeding education in the first phase of labor. A copy of the brochure will given to the pregnant women. In the early postpartum period, breastfeeding will encouraged practically and observed by the researchers. Participants' questions will answered. As a result, after the breastfeeding education, the mother will be evaluated with the breastfeeding efficiency scale and the maternal attachment scale.
  Interventions: Other: Group B
- Kontrol (No Intervention): No intervention will made to Group C by the researchers. Participants will benefit from the hospital's routine care and breastfeeding education services. As a result, postpartum mother will be evaluated with breastfeeding efficiency scale and maternal attachment scale.

INTERVENTIONS:
Behavioral: Group A — Skin-to-Skin Contact (SSC) contributes to mother-infant interaction and can increase breastfeeding success
  Other Names: Skin-to-skin Contact
  Arms: Skin-to-skin care
Other: Group B — education with a structured and expert opinion-based breastfeeding brochure
  Other Names: Breastfeeding education
  Arms: Breastfeeding Education

SUMMARY:
Objective: The study aimed to compare the effects of breastfeeding education and skin-to-skin contact on breastfeeding efficiency and maternal attachment.

Design: This study was planned as a three-group randomized controlled study. Setting and participants: This study will conduct with 92 women in a delivery room in Turkey between October 2021 and May 2022.

Methods: The study consists of continuous early skin-to-skin contact (SSC; Group A), breastfeeding education (Group B), and control groups (Group C). Group A received SSC education and Group B received structured breastfeeding education.

DETAILED DESCRIPTION:
Primiparous women in the latent phase will given detailed information about the study (purpose and benefits of the study) and the pregnant women will invited to the study. Pregnant women will assigned to one of three groups (1:1:1) as A, B, and C in the www.randomizer.org program. Prior to the interventions, the Mother-Infant Information Form and MAI will applied to the pregnant women. After the interventions, MAI and BBAT will applied at an appropriate time when the participants felt most comfortable and rested and their perceptions will clear (4-6 hours postpartum). Eventually, the study sample will composed of 93 pregnant women based on the CONSORT 2010 (http://www.consort-statement.org/) flow diagram: 31 participants in Group A, and 31 in the Groups B, C (Figure 1).

SSC (Group-A) Pregnant women will assigned to Group A will informed about SSC. SSC will ensured postpartum in a supported diagonal-flexion position continuously by the researchers for 45-120 minutes. Mothers in group A will also benefit from the hospital's routine breastfeeding education service.

Structured Breastfeeding Education Program (Group-B) Structured breastfeeding education material will prepared to increase breastfeeding awareness and level of knowledge. Opinions will received from 7 different experts for the education booklet and brochure. The material will revised based on expert opinions. A brochure and educational material will administered to 10 pregnant women before the study and the material will found to be understandable. The education booklet include breastfeeding techniques, the benefits of breast milk, the benefits of breastfeeding, solution suggestions for breastfeeding problems, lactation mechanism, and storage of breast milk. The breastfeeding brochure include educational texts, educators' contact information, and pictures.

Group B will receive face-to-face breastfeeding education in the first phase of labor. A copy of the brochure will given to the pregnant women. In the early postpartum period, breastfeeding will encouraged practically and observed by the researchers. Participants' questions will answered.

Control (Group-C) No intervention will made to Group C by the researchers. Participants benefite from the hospital's routine care and breastfeeding education services. Posttests will applied in a way that would not interrupt the routine care and education practices of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* were having a primiparous pregnancy,
* being open to cooperation,
* having a vaginal delivery,
* giving a single mature birth,
* having no communication problem

Exclusion Criteria:

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — postpartum women
Enrollment: 92 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Skin-to-skin contact | 6-8 hours
  Positive effect of skin-to-skin contact on maternal attachment and breastfeeding efficiency
Breastfeeding education | 6-8 hours
  positive effect of providing education with a structured and expert opinion-based breastfeeding brochure on maternal attachment and breastfeeding efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)